CLINICAL TRIAL: NCT03076983
Title: Assessment of the Capability of PulmoVista 500 to Continuously Monitor Changes of Ventilation Over Time
Status: Completed | Type: Observational
Sponsor: Drägerwerk AG & Co. KGaA (Industry)
Collaborators: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: PV500
Record Dates: First submitted 2017-02-22; First posted 2017-03-10 (Actual); Results first posted 2019-10-18 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Mechanical Ventilation; Single-lung Ventilation; ARDS; ALI - Acute Lung Injury; Weaning From Ventilator
Keywords: Ventilation Monitoring; Electrical Impedance Tomography
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU Patients: Patients currently on or scheduled for ventilator care in the intensive-care-unit (ICU)
  Interventions: Device: Lung Monitoring with EIT device (PulmoVista 500)
- OLV Patients: Patients scheduled for elective surgery receiving one-lung-ventilation (OLV)
  Interventions: Device: Lung Monitoring with EIT device (PulmoVista 500)

INTERVENTIONS:
Device: Lung Monitoring with EIT device (PulmoVista 500) — Patient's lungs will be monitored during clinical routine interventions with Dräger's EIT device (PulmoVista 500).
  No medical interventions to routine patient care required.

SUMMARY:
The results of this study will help to define the capability and reliability of PulmoVista 500 to detect changes in both global and regional ventilation.

ELIGIBILITY:
Inclusion Criteria

- The population included in the clinical study will be selected from a pool of patients undergoing respiratory support who are scheduled to have their ventilation settings changed.

As a subgroup, patients who are scheduled for surgeries that need one-lung-ventilation (OLV) will be enrolled to the study.

* Male and female patients at the age of 18 years or older
* On respiratory support in ICU care or scheduled for such ( e.g. postoperatively) or scheduled for surgery with OLV
* Patients of which the monitoring of ventilation distribution may be of clinical interest
* Patients being ventilated via an artificial airway with a mechanical ventilator that is compatible with PulmoVista 500
* Patients scheduled for changes in ventilation settings that may cause relevant changes in the ventilation
* Chest circumference between 70 and 150 cm
* Written informed consent to participate in the study provided by either the patient or the legal representative of the patient.

Exclusion Criteria

* Currently has a permanent or temporary pacemaker, implantable cardiac device (ICD) or other device emitting electrical energy
* a BMI ≥ 50
* tidal volume (VT) ≤ 200 mL
* Current uncontrolled body movements such as tics, tremors or seizures,
* Current wound dressings or infections on the chest that might interfere with the PulmoVista 500 electrode belt placement
* Women of child bearing potential whose pregnancy cannot be excluded based on a pregnancy test or other proven facts.
* Allergic to materials used in the electrode belt
* Participation of the patient in an interventional trial within the last four weeks before enrollment in this trial
* Evidence suggesting that the patient or his legal representative is not likely to follow the trial protocol (e.g. lacking compliance)
* Known infectious diseases that require isolation of patient (e.g. MRSA)
* Concomitant use of an air anti-decubitus medical mattress with dynamic inflation that cannot be deactivated during EIT measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit (ICU) patients, who are mechanically ventilated via an artificial airway (endotracheal tube or tracheostomy cannula) and who are expected to be subjected to major changes in their ventilator settings will be monitored with the PulmoVista 500 device before, during and after the changes. These changes in the ventilator settings should result in recognizable changes in the distribution of ventilation in the lungs.
  AND Patients who are scheduled for surgeries that require blocking of one bronchus
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Spieth, Prof.Dr. med., Principal Investigator — Universitätsklinikum Dresden; Oliver C Radke, Prof. Dr., Study Chair — Klinikum Bremerhaven-Reinkenheide gGmbH
Locations (3):
- Germany (3):
  - Klinikum Bremerhaven-Reinkenheide gGmbH, Bremerhaven
  - Universitätsklinik Dresden, Dresden
  - Medizinische Hochschule Hannover (MHH), Hanover

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ICU Patients: Patients currently on or scheduled for ventilator care in the intensive-care-unit (ICU)
  Lung Monitoring with EIT device (PulmoVista 500): Patient's lungs will be monitored during clinical routine interventions with Dräger's EIT device (PulmoVista 500).
  No medical interventions to routine patient care required.
- OLV Patients: Patients scheduled for elective surgery receiving one-lung-ventilation (OLV)
  Lung Monitoring with EIT device (PulmoVista 500): Patient's lungs will be monitored during clinical routine interventions with Dräger's EIT device (PulmoVista 500).
  No medical interventions to routine patient care required.
Period: Overall Study
Arm/Group | ICU Patients | OLV Patients
Started | 55 | 25
Completed | 55 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICU Patients | OLV Patients | Total
Number analyzed (Participants) | 55 | 25 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (13.8) | 59.1 (12.5) | 60.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 37 | 15 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 55 | 25 | 80
Region of Enrollment [Number; unit: participants]
  Germany | 55 | 25 | 80
Height [Mean (Standard Deviation); unit: Centimetre] | 172.02 (9.29) | 170.96 (10.69) | 171.69 (9.70)
Weight [Mean (Standard Deviation); unit: kilogram] | 79.75 (21.25) | 80.84 (15.68) | 80.09 (19.59)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.87 (6.33) | 27.62 (4.89) | 27.11 (5.90)

OUTCOME MEASURES:

1. Primary Outcome: Monitoring Capabilities of PulmoVista 500
Description: The cross-correlation between the volume curve of the ventilator and the global impedance curve of PulmoVista 500 was expressed by the cross-correlation coefficient R.
  The cross-correlation coefficient is a measure to quantify the relationship between the volume curve and the EIT curve.
  The correlation coefficient R can assume values between [-1, 1] to describe the relationship between the two curves, as is usual for a correlation.
  To calculate the correlation coefficient, a phase shift between the two curves was taken into account, so the cross-correlation between them was calculated.
  The phase shift or delay occurs when the signal from the fan is transmitted to the PulmoVista500.
  The cross-correlation coefficient is determined by calculating the correlation coefficient for the curves within a narrow range of Lags(-15 to 15 ) for each pair of curves and using the maximum value as the value of correlation coefficient (therefore it is called cross-correlation coefficient)
Time Frame: Day 1
Population: A Intention-to-Treat (ITT) collective was used as analysis population. The intention-to-treat collective comprises all patients for which both, the impedance waveforms and parallel to them volume waveforms have been generated during ventilation,so that the primary endpoint can be evaluated.
Measure: Mean (Standard Deviation); unit: correlation coefficient
Arm/Group | ICU Patients | OLV Patients
Number analyzed (Participants) | 54 | 25
correlation coefficient | 0.9692 (0.0627) | 0.9093 (0.1351)

2. Secondary Outcome: Detection of Changes in Regional Ventilation
Description: To assess the capability of PulmoVista 500 to detect changes in regional ventilation by evaluating the cross correlation between impedance waveforms derived from PulmoVista 500 and volume curves derived from ventilator during one-lung-ventilation.
Time Frame: Day 1
Population: For this secondary endpoint the cross-correlation between between impedance waveforms derived from PulmoVista 500 and volume curves derived from Ventilator was calculated only for patients which received one-lung-ventilation (OLV).
  Therefore no patients from the ICU patients Group were included into the analysis.
Measure: Mean (Standard Deviation); unit: correlation coefficient
Arm/Group | ICU Patients | OLV Patients
Number analyzed (Participants) | 0 | 25
correlation coefficient |  | 0.9093 (0.1351)

3. Secondary Outcome: Assess Changes of Tidal Volumes
Description: Assess that changes of tidal volumes induced by ventilator settings can be monitored by the "Trends view"
  To assess if the changes of tidal volumes induced by ventilator settings can be monitored by the "Trends view", the physician was asked to answer following question of a questionnaire:
  "Open the view "End-insp. trend" after the PEEP setting has been changed significantly (2 mbar or more). Set C1 at the lower and C2 at the higher PEEP level.
  Does the image Change: C2 minus C1 and/or the corresponding regional Tidal Variations show the expected redistribution of ventilation from ventral to dorsal?"
  Possible answers were: "No", "Yes" and "N/A"
Time Frame: Day 1
Population: This question is only applicable to the patient group of "ICU Patients" as no assessment of the changes of tidal volumes induced by ventilator settings was planned a priori for the "OLV" patient group.
Measure: Count of Participants; unit: Participants
Arm/Group | ICU Patients | OLV Patients
Number analyzed (Participants) | 55 | 0
Participants
  Answer:No | 3 |
  Answer: Yes | 49 |
  Answer: N/A | 3 |

4. Secondary Outcome: Assess Changes of the End-expiratory Lung Volumes
Description: Assess that changes of the end-expiratory lung volumes (induced by e.g. PEEP changes, recruitment and suctioning maneuvers) can be monitored by "dEELI trend view"
  To assess if the changes of the end-expiratory lung volumes (induced by e.g. PEEP changes, recruitment and suctioning maneuvers) can be monitored by "dEELI trend view", the physician was asked to answer following two question of a questionnaire:
  Question 1: "Open the view "dEELI trend" after the PEEP setting has been changed. Set C1 at the lower and C2 at the higher PEEP level. Does the image dEELI: C2 minus C1 show the expected increase of end-exp. lung volume in turquoise (light-blue)?"
  Question 2: "Open the view "dEELI trend" after lung suction has been conducted. Set C1 at a phase before and C2 during or immediately after the lung suction. Does the image dEELI: C2 minus C1 show the expected decrease of lung volume in orange color?"
  Possible answers for the both above mentioned questions were "No","Yes" or "N/A2
Time Frame: Day 1
Population: These two questions are only applicable to the patient group of "ICU Patients" as no assessment of the changes of the end-expiratory lung volume was planned a priori within the "OLV" patient group.
Measure: Count of Participants; unit: Participants
Arm/Group | ICU Patients | OLV Patients
Number analyzed (Participants) | 55 | 0
Participants
  Question 1: Answer: "No" | 1 |
  Question 1: Answer: "Yes" | 51 |
  Question 1: Answer: "N/A | 3 |
  Question 2: Answer: "No" | 0 |
  Question 2: Answer: "Yes" | 29 |
  Question 2: Answer: "N/A | 26 |

5. Secondary Outcome: Safety - Documentation of Any Safety Events
Description: Documentation of any safety events related to the use of PulmoVista 500
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | ICU Patients | OLV Patients
Number analyzed (Participants) | 55 | 25
Participants
  Subjects with any AE: no | 43 | 13
  Subjects with any AE: yes | 12 | 12
  Subjects with any ADE: no | 55 | 25
  Subjects with any ADE: yes | 0 | 0
  Subjects with any SAE: no | 48 | 24
  Subjects with any SAE: yes | 7 | 1

6. Secondary Outcome: Assessing the Use Specific Clinical Helpfulness of PulmoVista 500 by Particular Questionnaire. The Questions Which Were Asked Within the Questionaire Are Listed in the "Outcome Measure Description"
Description: "How easy is it to...
  Q1: ... identify within the Tidal Image, whether the right and the left lung are evenly ventilated?" Q2: ... quantify the regional ventilation distribution as expressed by the regional Parameters TV ROI 1 - TV ROI 4?" Q3: ... set the cursors to respective positions which allow you to compare ventilation distribution before and after the intervention?" Q4: ... detect increases and/or decreases of regional ventilation?" Q5: ... relate the regional ventilation distribution to and the corresponding parameters from the ventilator, which are displayed in the trend table to each other?" Q7: ... set the cursors to respective positions which allows you assessing lung volume changes induced by the intervention?" Q8: ... detect increases and/or decreases of regional lung volume?"
  "How useful is the clinical Information on...
  Q6: ... ventilation redistribution caused by this intervention?" Q9: ... regional lung volume changes caused by this intervention?"
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | ICU Patients | OLV Patients
Number analyzed (Participants) | 55 | 25
Participants
  Question 1: 1 = very difficult / not useful at all | 0 | 0
  Question 1: 2 | 0 | 0
  Question 1: 3 | 2 | 0
  Question 1: 4 | 1 | 0
  Question 1: 5 = very easy / very useful | 52 | 25
  Question 2: 1 = very difficult / not useful at all | 0 | 0
  Question 2: 2 | 0 | 0
  Question 2: 3 | 2 | 0
  Question 2: 4 | 3 | 3
  Question 2: 5 = very easy / very useful | 50 | 22
  Question 3: 1 = very difficult / not useful at all | 0 | 0
  Question 3: 2 | 0 | 0
  Question 3: 3 | 0 | 2
  Question 3: 4 | 0 | 2
  Question 3: 5 = very easy / very useful | 55 | 21
  Question 4: 1 = very difficult / not useful at all | 0 | 1
  Question 4: 2 | 0 | 1
  Question 4: 3 | 2 | 0
  Question 4: 4 | 2 | 3
  Question 4: 5 = very easy / very useful | 51 | 20
  Question 5: 1 = very difficult / not useful at all | 0 | 1
  Question 5: 2 | 0 | 1
  Question 5: 3 | 0 | 2
  Question 5: 4 | 2 | 9
  Question 5: 5 = very easy / very useful | 53 | 12
  Question 6: 1 = very difficult / not useful at all | 0 | 1
  Question 6: 2 | 0 | 1
  Question 6: 3 | 9 | 10
  Question 6: 4 | 11 | 11
  Question 6: 5 = very easy / very useful | 35 | 2
  Question 7: 1 = very difficult / not useful at all | 0 | 0
  Question 7: 2 | 0 | 1
  Question 7: 3 | 0 | 2
  Question 7: 4 | 0 | 5
  Question 7: 5 = very easy / very useful | 55 | 17
  Question 8: 1 = very difficult / not useful at all | 0 | 1
  Question 8: 2 | 0 | 2
  Question 8: 3 | 2 | 1
  Question 8: 4 | 3 | 5
  Question 8: 5 = very easy / very useful | 50 | 16
  Question 9: 1 = very difficult / not useful at all | 0 | 2
  Question 9: 2 | 0 | 2
  Question 9: 3 | 10 | 14
  Question 9: 4 | 10 | 6
  Question 9: 5 = very easy / very useful | 35 | 1

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected during the follow-up visit, which takes place once within 1-3 days period after the study day.
Arm/Group | ICU Patients | OLV Patients
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/25
Serious Adverse Events (participants affected / at risk) | 7/55 | 1/25
Other Adverse Events (participants affected / at risk) | 2/55 | 12/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICU Patients (N=55) | OLV Patients (N=25)
Post procedural swelling (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICU Patients (N=55) | OLV Patients (N=25)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 12 (12)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03076983/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT03076983/SAP_001.pdf